CLINICAL TRIAL: NCT05404776
Title: Tension Versus Tension-Free Foley Balloon for Cervical Ripening in Nulliparous Women Undergoing Induction of Labor: A Cluster Randomized Controlled Trial
Brief Title: Tension Versus Tension- Free Foley Balloon for Cervical Ripening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-0327
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Induced Vaginal Delivery
Keywords: Induced Vaginal Delivery; Cervical Ripening; Mechanical Cervical Ripening
MeSH Terms: interventions — Cervical Ripening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without tension (tension free) (Experimental): The study group will undergo induction of labor by placement of a transcervical Foley balloon. The balloon tubing will be left free of tension and will hang freely.
  Interventions: Other: Placement of Foley balloon for cervical ripening without tension.
- Tension (Active Comparator): The control group will undergo induction of labor by placement of a transcervical Foley balloon. The balloon tubing will be pulled to create tension and will then be taped to the patient's inner thigh.
  Interventions: Other: Placement of Foley balloon for cervical ripening with tension.

INTERVENTIONS:
Other: Placement of Foley balloon for cervical ripening with tension. — A Foley balloon will be placed for cervical ripening with tension.
  Arms: Tension
Other: Placement of Foley balloon for cervical ripening without tension. — A Foley balloon will be placed for cervical ripening without tension.
  Arms: Without tension (tension free)

SUMMARY:
Foley balloons are commonly used as a mechanical method of cervical ripening for induction of labor. Foley balloons may be placed either under tension or without tension (tension-free). The purpose of our study is to examine time to delivery in nulliparous women undergoing induction of labor who have a Foley balloon placed as a mechanical cervical dilator, assigned to either tension or without tension. The goal is to determine if there is a potential added benefit to placing the Foley balloon on tension as compared to no tension. Our hypothesis is that Foley balloon under tension for cervical ripening results in shorter time to vaginal delivery compared to Foley balloon placed without tension.

DETAILED DESCRIPTION:
This is a pragmatic cluster randomized clinical trial. The target population is nulliparous women who present for induction of labor at term. If there is a decision by the obstetric team to place a transcervical Foley dilator for cervical ripening in a prospective subject meeting inclusion criteria for the study, the obstetric provider will follow the weekly randomization sequence for study group (No Tension) or the control group (Tension) based on the assigned cluster for the entire unit for that week. Both study groups will receive standardized labor management as Foley balloon placed with tension and without tension are both considered standard of care at our institution.

The Tension standard of care (control group) will undergo induction of labor by placement of a transcervical Foley balloon, which is standard of care at our institution. The balloon tubing will be pulled to create tension and will then be taped to the patient's inner thigh.

The No Tension standard of care (study group) will undergo induction of labor by placement of a transcervical Foley balloon. The balloon tubing will be left free of tension and will hang freely.

Subjects in the control and study group will then undergo standard intrapartum care. The total participation time in the study will be considered terminated following delivery.

ELIGIBILITY:
Inclusion Criteria:

* Term induction of labor
* Nulliparous
* Vertex
* Singleton
* Plan for Foley balloon placement by the managing obstetrics team
* Cervical exam less than 3 cm dilated and less than or equal to 60% effaced

Exclusion Criteria:

* Patient unwilling or unable to provide verbal consent
* Fetal demise or major congenital anomaly
* Preterm (<37 0/7weeks)
* Multiple gestation
* Previous uterine surgery
* Abnormal placentation
* Malpresentation
* Magnesium infusion for preeclampsia with severe features
* Prelabor rupture of membranes
* Fetal growth restriction
* Non-reassuring fetal heart rate tracing prior to inclusion

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meagan V Benson, DO, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Study records will be kept confidential as required by law. No IPD will be shared outside of UTMB. Identifiers will not be disclosed outside of the University of Texas Medical Branch (UTMB). The data collected will be kept on a password-secured UTMB computer. An encrypted USB flash drive will be used to transfer data. During analysis of the data, all identifiers will be deleted.

REFERENCES:
- [Background] Adhikari EH, Nelson DB, McIntire DD, Leveno KJ. Foley Bulb Added to an Oral Misoprostol Induction Protocol: A Cluster Randomized Trial. Obstet Gynecol. 2020 Nov;136(5):953-961. doi: 10.1097/AOG.0000000000004123. PMID 33030881
- [Background] Connolly KA, Kohari KS, Factor SH, Rekawek P, Miller MR, Smilen BS, Stone JL, Bianco AT. A Randomized Trial of Foley Balloon Induction of Labor Trial in Multiparas (FIAT-M). Am J Perinatol. 2017 Sep;34(11):1108-1114. doi: 10.1055/s-0037-1603994. Epub 2017 Jun 26. No abstract available. PMID 28651258
- [Background] Connolly KA, Kohari KS, Rekawek P, Smilen BS, Miller MR, Moshier E, Factor SH, Stone JL, Bianco AT. A randomized trial of Foley balloon induction of labor trial in nulliparas (FIAT-N). Am J Obstet Gynecol. 2016 Sep;215(3):392.e1-6. doi: 10.1016/j.ajog.2016.03.034. Epub 2016 Mar 24. PMID 27018464
- [Background] Fruhman G, Gavard JA, Amon E, Flick KV, Miller C, Gross GA. Tension compared to no tension on a Foley transcervical catheter for cervical ripening: a randomized controlled trial. Am J Obstet Gynecol. 2017 Jan;216(1):67.e1-67.e9. doi: 10.1016/j.ajog.2016.09.082. Epub 2016 Sep 15. PMID 27640940
- [Background] El Khouly NI. A prospective randomized trial comparing Foley catheter, oxytocin, and combination Foley catheter-oxytocin for labour induction with unfavourable cervix. J Obstet Gynaecol. 2017 Apr;37(3):309-314. doi: 10.1080/01443615.2016.1239075. Epub 2016 Dec 6. PMID 27922285
- [Background] Grobman WA, Rice MM, Reddy UM, Tita ATN, Silver RM, Mallett G, Hill K, Thom EA, El-Sayed YY, Perez-Delboy A, Rouse DJ, Saade GR, Boggess KA, Chauhan SP, Iams JD, Chien EK, Casey BM, Gibbs RS, Srinivas SK, Swamy GK, Simhan HN, Macones GA; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Labor Induction versus Expectant Management in Low-Risk Nulliparous Women. N Engl J Med. 2018 Aug 9;379(6):513-523. doi: 10.1056/NEJMoa1800566. PMID 30089070
- [Background] Kuhlmann MJ, Spencer N, Garcia-Jasso C, Singh P, Abdelwahab M, Vaughn M, Marshall K, Prasad N, Soulsby-Monroy R, Saade GR, Saad AF. Foley Bulb Insertion by Blind Placement Compared With Direct Visualization: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):139-145. doi: 10.1097/AOG.0000000000004182. PMID 33278290
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] McMaster K, Sanchez-Ramos L, Kaunitz AM. Evaluation of a Transcervical Foley Catheter as a Source of Infection: A Systematic Review and Meta-analysis. Obstet Gynecol. 2015 Sep;126(3):539-551. doi: 10.1097/AOG.0000000000001002. PMID 26244535
- [Background] Embrey MP, Mollison BG. The unfavourable cervix and induction of labour using a cervical balloon. J Obstet Gynaecol Br Commonw. 1967 Feb;74(1):44-8. doi: 10.1111/j.1471-0528.1967.tb03931.x. No abstract available. PMID 6018096
- [Background] Jozwiak M, Bloemenkamp KW, Kelly AJ, Mol BW, Irion O, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2012 Mar 14;(3):CD001233. doi: 10.1002/14651858.CD001233.pub2. PMID 22419277
- [Background] Schoen CN, Grant G, Berghella V, Hoffman MK, Sciscione A. Intracervical Foley Catheter With and Without Oxytocin for Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2017 Jun;129(6):1046-1053. doi: 10.1097/AOG.0000000000002032. PMID 28486381
- [Background] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515
- [Derived] Benson M, Younes L, Watson A, Saade GR, Saad AF. Applying Tension to the Transcervical Foley Balloon and Delivery Times in Term Nulliparous Women Undergoing Induction of Labor: A Randomized Controlled Trial. Obstet Gynecol. 2024 May 1;143(5):670-676. doi: 10.1097/AOG.0000000000005546. Epub 2024 Feb 29. PMID 38422505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The intervention is assigned at the cluster (weekly) level; the total number of participants enrolled will be reported as a single total and not separated by clusters.
Groups:
- Without Tension (Tension Free): A Foley balloon is introduced into the cervix either manually or under direct visualization, but the foley will not be taped or under tension.
  Placement of Foley balloon for cervical ripening without tension. A Foley balloon will be placed for cervical ripening without tension.
- Tension: The control group will undergo induction of labor by placement of a transcervical Foley balloon. The balloon tubing will be pulled to create tension and will then be taped to the patient's inner thigh.
  Placement of Foley balloon for cervical ripening with tension. A Foley balloon will be placed for cervical ripening with tension.
Period: Overall Study
Arm/Group | Without Tension (Tension Free) | Tension
Started | 141 | 138
Completed | 141 | 138
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Without Tension (Tension Free) | Tension | Total
Number analyzed (Participants) | 141 | 138 | 279
Age, Continuous [Median (Full Range); unit: years] | 23 [18 to 39] | 22 [18 to 42] | 22 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 138 | 279
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 94 | 88 | 182
  Not Hispanic or Latino | 47 | 50 | 97
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 115 | 122 | 237
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 141 | 138 | 279

OUTCOME MEASURES:

1. Primary Outcome: Time to Vaginal Delivery
Description: Time to vaginal delivery measured from time of initial Foley balloon placement to delivery
Time Frame: Foley bulb placement to vaginal delivery, up to 24 Hours
Measure: Median (Full Range); unit: minutes
Arm/Group | Without Tension (Tension Free) | Tension
Number analyzed (Participants) | 99 | 91
minutes | 1608 [430 to 3438] | 1595.5 [507 to 3323]

2. Secondary Outcome: Number of Participants That Requested Analgesia Following Placement of the Foley Balloon
Description: Request for IV pain medications or epidural following placement of Foley balloon
Time Frame: Placement of Foley balloon until removal of Foley balloon in minutes (up to 12 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Without Tension (Tension Free) | Tension
Number analyzed (Participants) | 141 | 138
Participants | 119 | 114

3. Secondary Outcome: Number of Participants That Had a Primary Cesarean Delivery
Description: Number of participants that had a primary cesarean delivery
Time Frame: Placement of Foley balloon until cesarean delivery, up to 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Without Tension (Tension Free) | Tension
Number analyzed (Participants) | 141 | 138
Participants | 42 | 47

4. Secondary Outcome: Number of Participants With Chorioamnionitis
Description: Number of participants with chorioamnionitis
Time Frame: Placement of Foley balloon until delivery, up to 24 Hours
Measure: Count of Participants; unit: Participants
Arm/Group | Without Tension (Tension Free) | Tension
Number analyzed (Participants) | 141 | 138
Participants | 40 | 48

5. Other Pre Specified Outcome: Number of Participants With Postpartum Hemorrhage
Description: Number of participants with postpartum hemorrhage
Time Frame: Placement of Foley balloon until 24 hours postpartum
Population: Outcome measure not assessed
Arm/Group | Without Tension (Tension Free) | Tension
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Without Tension (Tension Free) | Tension
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/138
Other Adverse Events (participants affected / at risk) | 0/141 | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/76/NCT05404776/Prot_SAP_000.pdf